CLINICAL TRIAL: NCT03694444
Title: A Phase 2a Clinical Trial to Assess the Safety and Efficacy of C3 Inhibitor AMY-101, in Adults With Gingivitis
Brief Title: A Study of the C3 Complement Inhibitor AMY-101 in Adults With Gingivitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amyndas Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMY-101/perio1
Record Dates: First submitted 2018-09-23; First posted 2018-10-03 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — AMY-101; Water; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMY-101 treatment (Active Comparator): Subjects who meet inclusion criteria will be enrolled in the study and sites will be randomized to treatment groups (AMY-101 or placebo) in split mouth design. In the AMY-101 treatment arm after clinical assessments and sample collection at baseline, test treatments will be administered to each of the interproximal papilla and will be repeated on Day 7 and 14.
  Interventions: Drug: AMY-101
- Placebo (Placebo Comparator): Subjects who meet inclusion criteria will be enrolled in the study and sites will be randomized to treatment groups (AMY-101 or placebo) in split mouth design. In the placebo arm, after clinical assessments and sample collection at baseline, placebo treatments will be administered to each of the interproximal papilla and will be repeated on Day 7 and 14.
  Interventions: Other: Water for injection

INTERVENTIONS:
Drug: AMY-101 — C3 complement inhibitor
  Arms: AMY-101 treatment
Other: Water for injection — Placebo
  Arms: Placebo

SUMMARY:
A Phase 2a Clinical Trial to Assess the Safety and Efficacy of Complement 3 Inhibitor Analog, AMY-101, in Adults with gingivitis.

The study is a 3-month randomized, double-blind, split-mouth study of adults with existing chronic periodontal inflammation determined by the level of gingival index and bleeding on probing. The primary endpoint of change in gingival index will be evaluated at 21, 28 and 90 days after initial treatment (baseline treatment). Subjects will also be followed at Day 3, 7, 14, 21, 28 and 90 for safety evaluations. Change in bleeding on probing plaque index, pocket depth, clinical attachment level and GCF levels of pro-inflammatory cytokines and complement factors will be assessed as secondary outcome measures. Composition of subgingival biofilm will be assessed as an exploratory endpoint.

Subjects who meet inclusion criteria will be enrolled in the study and sites will be randomized to treatment groups (AMY-101 or placebo) in split mouth design. After clinical assessments and sample collection at baseline, both test and placebo treatments will be administered to each of the interproximal papilla and will be repeated on Day 7 and 14.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Age 18-65 years old.
4. Equal to or greater than 18 natural teeth present (excluding third molars).
5. Generalized periodontal inflammation determined by modified gingival index and percent bleeding on probing (MGI≥2.0, BOP ≥ 40%).
6. In good general health as evidenced by medical history.
7. For women of reproductive potential, use of licensed hormonal contraception or barrier methods or abstinence for at least 1 month prior to screening and agreement to use such a method during study participation.
8. For men of reproductive potential, agreement to use condoms or other methods to ensure effective contraception with partner.

Exclusion Criteria:

1. Presence of orthodontic appliances (including fixed lingual retainer).
2. A soft or hard tissue tumor of the oral cavity.
3. Carious lesions requiring immediate treatment.
4. Participation in any other clinical study within 30 days of screening or during the study.
5. Antibiotic therapy within the last 30 days.
6. Chronic use (≥3 times/week) of anti-inflammatory medications [e.g., non-steroidal anti-inflammatory drugs (NSAIDs), steroids]. Low dose (<325 mg) aspirin is allowed.
7. Immune compromised subjects (e.g., subjects with HIV infection, neutropenia, complement deficiency, etc.).
8. Any medical history or any concomitant medication that might affect the assessment of the study treatment or periodontal tissues, such as diabetes (irrespective of level of control), rheumatoid arthritis, Crohn's disease, nifedipine, phenytoin (Dilantin), anticoagulant medications (e.g., warfarin [Coumadin] etc.), ongoing cancer treatment either with radiation or chemotherapy.
9. Involvement in the planning or conduct of the study.
10. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or interfere with interpretation of the subject's study results.
11. Pregnancy or lactation.
12. Uncontrolled chronic diseases (e.g., kidney disease, COPD, pulmonary fibrosis, Hepatitis C)
13. Autoimmune disorders (Down's Syndrome, Sjogren's Disease, Psoriasis, Chediak-Higashi Syndrome)
14. Conditions requiring antibiotic prophylaxis.
15. Periodontal therapy within the past one year.
16. Gross tooth decay, as determined by the investigator.
17. Periodontal or dental abscesses.
18. Root fragments, pericoronitis, endo-perio lesions.
19. Use of cigarettes or other tobacco products (including e-cigarette or recreational drug use) within 1 year before the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Change in mean gingival index (MGI) | Assessed at 28 days after initial treatment

SECONDARY OUTCOMES:
Gingival inflammation | Assessed at baseline and Days 3, 7, 14, 21, and 28.
Ulceration in the oral cavity | Assessed at baseline and Days 3, 7, 14, 21, and 28.
Oral infections | Assessed at baseline and Days 3, 7, 14, 21, and 28.
Changes in mean gingival index | Assessed at Days 21 and 90
Changes in mean bleeding on probing (BOP) | Assessed at baseline and 21, 28 and 90 days
Changes in mean probing depth (PD) | Assessed at baseline and 21, 28 and 90 days
Number of sites with PD greater or equal to 5 mm | Assessed at baseline and 21, 28 and 90 days
Changes in mean clinical attachment level (CAL) | Assessed at baseline and 21, 28 and 90 days
Changes in plaque index (PI) | Assessed at baseline and 21, 28 and 90 days
Levels of gingival crevicular fluid (GCF) | Assessed at baseline and 21, 28 and 90 days
Levels of proinflammatory mediators in the GCF | Assessed at baseline and 21, 28 and 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Forsyth Institute, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Hasturk H, Hajishengallis G; Forsyth Institute Center for Clinical and Translational Research staff; Lambris JD, Mastellos DC, Yancopoulou D. Phase IIa clinical trial of complement C3 inhibitor AMY-101 in adults with periodontal inflammation. J Clin Invest. 2021 Dec 1;131(23):e152973. doi: 10.1172/JCI152973. PMID 34618684
- [Derived] Hajishengallis G, Hasturk H, Lambris JD; Contributing authors. C3-targeted therapy in periodontal disease: moving closer to the clinic. Trends Immunol. 2021 Oct;42(10):856-864. doi: 10.1016/j.it.2021.08.001. Epub 2021 Sep 2. PMID 34483038